CLINICAL TRIAL: NCT03657069
Title: A Pilot Study of Applying New Device Technologies for Tissue Expander/Implant-Based Breast Reconstruction (Blossom Syringe Assist Device)
Brief Title: Blossom Smart Expander Technology in Breast Reconstruction in Participants With Breast Cancer Undergoing Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Dung Nguyen, Clinical Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-44367; NCI-2018-01702 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRS0088 (Other: OnCore)
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-04

CONDITIONS: Breast Carcinoma; Breast Disorder
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Supportive care (Blossom Smart Expander Technology) (Experimental): After mastectomy, participants undergo 2-staged IBR with the Blossom Smart Expander Technology comprising of the Blossom syringe assist device connected to the Mentor SPECTRUM adjustable saline breast implant.
  Interventions: Device: Blossom; Other: Breast-Q -Reconstruction module (preoperative) version 2.0 satisfaction with breasts questionnaire

INTERVENTIONS:
Device: Blossom — Undergo Implant Breast Reconstruction (IBR) with the Blossom Smart Expander Technology
  Other Names: Blossom Smart Expander Technology (Syringe Assist Device)
Other: Breast-Q -Reconstruction module (preoperative) version 2.0 satisfaction with breasts questionnaire — Ancillary studies

SUMMARY:
This phase 1 trial studies how well Blossom Smart Expander Technology works in breast reconstruction in participants with breast cancer undergoing mastectomy. Blossom Smart Expander Technology allows for slow and continuous injection of small amounts of saline, from an external pouch and based on precise pressure and volume measurements, into breast expander implants. It may help in achieving the same reconstructive goals as conventional tissue expansion in a shorter period of time and while avoiding frequent injections through the skin, which cause patient discomfort and require many clinic visits.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the clinical effectiveness of the application of Blossom Smart Expander Technology in 2-staged tissue expander/implant-based breast reconstruction.

SECONDARY OBJECTIVES:

I. Patient satisfaction. II. Patient self-reported pain. III. Incidence of complications.

OUTLINE:

After mastectomy, participants undergo 2-staged implant-based breast reconstruction (IBR) with the Blossom Smart Expander Technology comprising of the Blossom syringe assist device connected to the Mentor SPECTRUM adjustable saline breast implant.

After completion of study treatment, participants are followed up at 1 week and then every week or every month thereafter for up to 12 months

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer or reason for prophylactic mastectomy (e.g., BRCA mutation and/or strong family history of breast cancer), both unilateral or bilateral mastectomy
* No prior breast surgery (excluding biopsy and lumpectomy) or breast radiation
* Ability to understand and the willingness to sign a written informed consent document
* No life expectancy restrictions
* Eastern Cooperative Oncology Group (ECOG) or Karnofsky performance status will not be employed
* No requirements for organ and marrow function

Exclusion Criteria:

* Recent steroid use
* No major medical comorbidities (defined as American Society of Anesthesiologists [ASA] III or greater)
* No connective tissue disorder
* Prior breast surgery, excluding biopsy and lumpectomy
* History of or plan for breast radiation
* Pregnancy and nursing patients will be excluded from the study
* No restrictions regarding use of other investigational agents
* No exclusion criteria related to history of allergic reactions
* No exclusion criteria relating to concomitant medications or substances that have the potential to affect the activity or pharmacokinetics of the study agent
* No other agent-specific exclusion criteria
* No exclusion of cancer survivors or those who are human immunodeficiency virus (HIV)-positive

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung Nguyen, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: breasts
Groups:
- Supportive Care (Blossom Smart Expander Technology): After mastectomy, participants undergo 2-staged IBR with the Blossom Smart Expander Technology comprised of the Blossom syringe assist device connected to the Mentor SPECTRUM adjustable saline breast implant.
Period: Overall Study
Arm/Group | Supportive Care (Blossom Smart Expander Technology)
Started | 11; 22 breasts
Completed | 11; 22 breasts
Not Completed | 0; 0 breasts

BASELINE CHARACTERISTICS:
Groups:
- Supportive Care (Blossom Smart Expander Technology): After mastectomy, participants undergo 2-staged IBR with the Blossom Smart Expander Technology.
Arm/Group | Supportive Care (Blossom Smart Expander Technology)
Number analyzed (Participants) | 11
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [35 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5
  Asian | 3
  Hispanic | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 20.6 [18.8 to 24.5]

OUTCOME MEASURES:

1. Primary Outcome: Time to Full Expansion Defined as Number of Days Until Desired Breast Tissue Expansion Volume is Achieved
Description: Measured by calculating the number of days from expander placement to achievement of desired expansion volume. Data were collected on a weekly basis until completion of breast expansion along with stabilization of surgical scars and percutaneous drain removal.
Time Frame: Assessed weekly for up to 12 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Supportive Care (Blossom Smart Expander Technology)
Number analyzed (Participants) | 11
days | 13 [8 to 18]

2. Secondary Outcome: BREAST-Q Reconstruction Module Version 2.0 Patient Satisfaction Score
Description: Defined as patient satisfaction with expansion process. Score range: 1 to 5 (5=very satisfied, 4=somewhat satisfied, 3=neutral, 2=somewhat dissatisfied, 1=very dissatisfied). Data were collected on a weekly basis until completion of breast expansion along with stabilization of surgical scars and percutaneous drain removal. Scores were averaged to create an overall score.
Time Frame: Assessed weekly for up to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care (Blossom Smart Expander Technology)
Number analyzed (Participants) | 11
score on a scale | 4.8 (0.39)

3. Secondary Outcome: Number of Participants With Major Complications Associated With Tissue Expansion Process
Description: Anticipated complications include Expander Extrusion, Wound Breakdown, and/or Infection. Data were collected on a weekly basis until completion of breast expansion along with stabilization of surgical scars and percutaneous drain removal.
Time Frame: Assessed weekly for up to 12 weeks
Measure: Count of Units; unit: breasts
Units Other Than Participants: breasts
Arm/Group | Supportive Care (Blossom Smart Expander Technology)
Number analyzed (Participants) | 11
Number analyzed (breasts) | 22
breasts
  Infection requiring IV antibiotics | 0
  Infection resulting in TE removal | 1
  Any other issues requiring surgical intervention | 0

4. Secondary Outcome: Number of Participants With Minor Complications Associated With Tissue Expansion Process
Description: as for outcome 3
Time Frame: Assessed weekly for up to 12 weeks
Measure: Count of Units; unit: breasts
Units Other Than Participants: breasts
Arm/Group | Supportive Care (Blossom Smart Expander Technology)
Number analyzed (Participants) | 11
Number analyzed (breasts) | 22
breasts
  Seroma | 1
  Hematoma | 0
  Infection resolved with oral antibiotics | 0
  Dehiscence, skin breakdown, etc. | 0

5. Secondary Outcome: Number of Participants With Device Malfunction Associated With Tissue Expansion Process
Description: Data were collected on a weekly basis until completion of breast expansion along with stabilization of surgical scars and percutaneous drain removal.
Time Frame: Assessed weekly for up to 12 weeks
Measure: Count of Units; unit: breasts
Units Other Than Participants: breasts
Arm/Group | Supportive Care (Blossom Smart Expander Technology)
Number analyzed (Participants) | 11
Number analyzed (breasts) | 22
breasts | 0

6. Secondary Outcome: Pain Score
Description: Self-reported pain associated with expansion process. Patients will be asked to rank pain level on a scale of 0 to 10, with 0 being the least pain and 10 being the most pain. Data were collected on a weekly basis until completion of breast expansion along with stabilization of surgical scars and percutaneous drain removal. Scores were averaged to create an overall score.
Time Frame: Assessed weekly for up to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care (Blossom Smart Expander Technology)
Number analyzed (Participants) | 11
score on a scale | 1.27 (1.35)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Supportive Care (Blossom Smart Expander Technology)
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Supportive Care (Blossom Smart Expander Technology) (N=11)
Infection (Infections and infestations) | 1 — Infection resulting TE removal
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Supportive Care (Blossom Smart Expander Technology) (N=11)
Seroma (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT03657069/Prot_SAP_000.pdf